CLINICAL TRIAL: NCT05906745
Title: Guideline Directed Medical Therapy (GDMT) Optimization and Adherence Longitudinal Study for Heart Failure. (GOALS-HF)
Brief Title: Guideline Directed Medical Therapy (GDMT) Optimization and Adherence Longitudinal Study for Heart Failure.
Acronym: GOALS-HF
Status: Completed | Type: Observational
Sponsor: Tricog Health Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TR001
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multicenter, non-randomized prospective longitudinal study to evaluate the feasibility of Tricog's Remote platform for Guideline Directed Medical Therapy (GDMT) titration and remote patient monitoring among patients with Heart Failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Recent hospitalization (within 4 weeks of enrollment) for HF with IV diuretic use
3. Echocardiographic data with EF measurements available in the last 6 months and after HF diagnosis
4. Established outpatient care at the participating sites
5. Eligible to receive at least 2 of the 4 GDMT classes (ACEi/ARB/ARNi, Beta-blockers, MRA, and SGLT2i) for HFrEF and HFmrEF and at least one of the three (ARB/ARNI, MRA, SGLT2i) for HFpEF
6. Not on Target GDMT for all the eligible GDMT classes
7. >12 months of expected survival
8. Comfortable with spoken and written English communication
9. Access to Apple Watch-compatible iPhone

Exclusion Criteria:

1. Under consideration for or recipient of advanced heart failure therapies (LVAD, Transplant)
2. Current or anticipated use of home intravenous inotrope therapy.
3. Unwilling or unable to perform all study related procedures (wear watch, take measurements and maintain daily logs)
4. Post-discharge placement in nursing, rehabilitation, or long-term care facility
5. Planned (within next 6 months) surgery
6. Inability to provide written consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults hospitalized for decompensated heart failure or in the post-discharge period following a heart failure hospitalization will be eligible for enrollment. Participants that meet eligibility criteria will be enrolled consecutively.
  Heart Failure with preserved ejection Fraction (HFpEF) will be defined by EF ≥ 50% at the time of HF diagnosis. Heart Failure with reduced ejection fraction (HFrEF) will be defined by EF <40%, and patients with EF between 40-49% will be identified as Heart Failure with mildly reduced EF (HFmrEF).
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
NT-ProBNP | Baseline, week 2, 1-month follow-up, week 8, 3-month follow-up, week 16, week 20, 6-month follow-up
  Serum level of N-terminal pro B-type natriuretic peptide

SECONDARY OUTCOMES:
HF Hospitalizations | 3-month, and 6-month follow-up
  Hospitalizations for heart failure
6-min walk distance | Baseline, 1-month follow-up, 3-month, and 6-month follow-up
  Six-minute walk test distance in meters
KCCQ Overall Summary Score | The survey will be assessed at baseline, 1-month, 3-month, and 6-month follow-up.
  The KCCQ summary score ranges from 0 to 100, where higher scores indicate better quality of life.
Atrial Fibrillation Anticoagulation Utilization | Baseline, 3-month, and 6-month
  Percentage of participants with atrial fibrillation indicated for anticoagulation that are on systemic anticoagulation.
HFpEF Medication Utilization | Baseline, 1-month follow-up, 3-month, and 6-month follow-up
  Percentage of participants on all three classes (ACEi/ARB/ARNI or MRA or SGLT2i)
composite modified HF Collaboratory GDMT score | Baseline, 1-month follow-up, 3-month, and 6-month follow-up
  2 points for optimal dosing of each medication class (beta-blockers, ACEi/ARB/ARNI, MRA, SGLT2i) and 1 point for suboptimal beta-blocker or ACEi/ARB dosing, expressed as a percentage of maximum possible points.
Changes in Diuretic Dose | 3-month, 6-month
  The number of days on higher than baseline dose of diuretic

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
- India (2):
  - Manipal Hospital, Bengaluru, Karnataka
  - Sakra World Hospital, Bengaluru, Karnataka

IPD SHARING:
Plan to Share IPD: No